CLINICAL TRIAL: NCT01179217
Title: A PHASE III, PROSPECTIVE, RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED, PARALLEL-GROUP, MULTICENTER STUDY OF L GLUTAMINE THERAPY FOR SICKLE CELL ANEMIA AND SICKLE ß0-THALASSEMIA
Brief Title: A Phase III Safety and Efficacy Study of L-Glutamine to Treat Sickle Cell Disease or Sickle βo-thalassemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Emmaus Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GLUSCC09-01
Record Dates: First submitted 2010-05-21; First posted 2010-08-11 (Estimated); Results first posted 2017-08-10 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2017-07

CONDITIONS: Sickle Cell Anemia; Sickle ß0-Thalassemia
Keywords: Sickle Cell Anemia; Sickle Cell Pain Crises; Painful Crises; Sickle Cell Pain; Vaso-occlusive Crises
MeSH Terms: conditions — Anemia, Sickle Cell; Vaso-Occlusive Crises | interventions — Glutamine; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- L-glutamine (Experimental): Patients will be randomized to receive investigational product, L-Glutamine.
  Interventions: Drug: L-glutamine
- 100% maltodextrin (Placebo Comparator): Patients will be randomized to receive Placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: L-glutamine — 0.3 g/kg of L-glutamine will be administered twice a day orally to each patient for 48 weeks. The dosage will be in increments of 5 grams based on weight. The upper limit for daily dose of study medication will be set at 30 grams. Patients will be given verbal and written instructions for self-administration of the study medication at the Baseline visit. The powder can be mixed with water or most non-heated beverages other than alcohol, or can be mixed with most non-heated foods such as yogurt, applesauce, or cereal for administration. Mixing L-glutamine with soda or highly acidic juices (such as grapefruit juice or lemonade) is not recommended.
  Other Names: oral L-glutamine
  Arms: L-glutamine
Drug: Placebo — 0.3 g/kg of placebo (100% maltodextrin) will be administered twice a day orally to each patient for 48 weeks. The dosage will be in increments of 5 grams based on weight. The upper limit for daily dose of study medication will be set at 30 grams. Patients will be given verbal and written instructions for self-administration of the study medication at the Baseline visit. The powder can be mixed with water or most non-heated beverages other than alcohol, or can be mixed with most non-heated foods such as yogurt, applesauce, or cereal for administration.
  Other Names: Maltodextrin
  Arms: 100% maltodextrin

SUMMARY:
The purpose of this research is to evaluate the effects of L-glutamine as a therapy for Sickle Cell Anemia or Sickle ß0 Thalassemia as evaluated by the number of occurrences of sickle cell crises.

DETAILED DESCRIPTION:
Primary objective:

To evaluate the efficacy of oral L-glutamine as a therapy for sickle cell anemia and sickle ß0-thalassemia as evaluated by the number of occurrences of sickle cell crises.

Secondary objectives:

To assess the effect of oral L-glutamine on: (a) frequency of hospitalizations for sickle cell pain; (b) frequency of emergency room/medical facility visits for sickle cell pain; and (c) hematological parameters (hemoglobin, hematocrit, and reticulocyte count); and to assess the safety of L-glutamine as a therapy for sickle cell anemia as evaluated by adverse events, laboratory parameters, and vital signs.

Methodology:

This was a 2:1 randomized, double-blind, placebo-controlled, parallel-group, multicenter study in patients with sickle cell anemia and sickle ß0-thalassemia who were at least 5 years old. Informed consent was obtained up to four weeks prior to Week 0 (Baseline). Screening procedures were performed anytime between the date of consent and Week 0, as long as all eligibility criteria had been confirmed prior to Week 0. At Week 0, patients were randomized (to L-glutamine or placebo) and underwent 48 weeks of treatment (orally BID), with dose calculated according to patient weight. Patient clinic visits occurred every 4 weeks, and phone calls took place between visits to monitor compliance. After 48 weeks of treatment, the dose was tapered to 0 within 3 weeks. A final evaluation visit occurred 2 weeks after last dose for a total of 53 weeks on study.

ELIGIBILITY:
Inclusion Criteria:

* Patient is at least five years of age.
* Patient has been diagnosed with sickle cell anemia or sickle ß°-thalassemia (documented by hemoglobin electrophoresis).
* Patient has had at least two documented episodes of sickle cell crises within 12 months of the screening visit.
* If the patient has been treated with an anti-sickling agent within three months of the screening visit, the therapy must have been continuous for at least three months with the intent to continue for the duration of the study.
* Patient or the patient's legally authorized representative has given written informed consent.
* If the patient is a female of child-bearing potential, she agrees to avoid pregnancy during the study and is willing and agrees to practice a recognized form of birth control during the course of the study (e.g. barrier, birth control pills, abstinence).

Exclusion Criteria:

* Patient has a significant medical condition that required hospitalization (other than sickle cell crisis) within two months of the screening visit.
* Patient has prothrombin time INR > 2.0.
* Patient has serum albumin < 3.0 g/dl.
* Patient has received any blood products within three weeks of the Screening Visit.
* Patient has uncontrolled liver disease or renal insufficiency.
* Patient is pregnant or lactating or has the intention of becoming pregnant during the study (if female and of child-bearing potential).
* Patient is currently taking or has been treated with any form of glutamine supplement within 30 days of the screening visit.
* Patient has been treated with an experimental anti-sickling medication/ treatment within 30 days of the screening visit (with the exception of hydroxyurea in pediatric patients).
* Patient is currently taking or has been treated with an investigational drug within 30 days of the screening visit (with the exception of hydroxyurea in pediatric patients).
* Patient is currently enrolled in an investigational drug or device study and/or has participated in such a study within 30 days of the screening visit.
* There are factors that would, in the judgment of the investigator, make it difficult for the patient to comply with the requirements of the study.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2010-05; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yutaka Niihara, MD, MPH, Study Director — Chairman and CEO
Locations (31):
- United States (31):
  - University of South Alabama Medical Center, Mobile, Alabama
  - Phoenix Children's Hospital Center for Cancer and Blood Disorders, Phoenix, Arizona
  - Kaiser Permanente, Inglewood, California
  - Children's Hospital & Research Center at Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Harbor-UCLA Medical Center, Torrance, California
  - University of Denver School of Medicine Sickle Cell Treatment & Research Center, Aurora, Colorado
  - Howard University Hospital & Howard University, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - Children's Healthcare of Atlanta at Egleston/Emory University, Atlanta, Georgia
  - University of Illinois at Chicago, Chicago, Illinois
  - University of Louisville School of Medicine, Louisville, Kentucky
  - Sickle Cell Center of S. Louisiana, Tulane University School of Medicine, New Orleans, Louisiana
  - Johns Hopkins University, Baltimore, Maryland
  - Boston University Medical Center, Boston, Massachusetts
  - Children's Hospital of Michigan, Detroit, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Children's Specialty Center of Nevada, Las Vegas, Nevada
  - Comprehensive Cancer Center of Nevada, Las Vegas, Nevada
  - Cooper University Hospital, Camden, New Jersey
  - The Brooklyn Hospital Center, Brooklyn, New York
  - SUNY - Downstate Medical Center, Brooklyn, New York
  - Brookdale University Hospital and Medical Center, Brooklyn, New York
  - New York Methodist Hospital - SC/Thalassemia Program, Brooklyn, New York
  - Interfaith Medical Center, Brooklyn, New York
  - Bronx Lebanon Hospital, The Bronx, New York
  - Presbyterian Blume Pediatric Hematology-Oncology Clinic, Charlotte, North Carolina
  - University of Tennessee Cancer Institute, Memphis, Tennessee
  - Virginia Commonwealth University, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bolarinwa AB, Oduwole O, Okebe J, Ogbenna AA, Otokiti OE, Olatinwo AT. Antioxidant supplementation for sickle cell disease. Cochrane Database Syst Rev. 2024 May 22;5(5):CD013590. doi: 10.1002/14651858.CD013590.pub2. PMID 38775255
- [Derived] Niihara Y, Miller ST, Kanter J, Lanzkron S, Smith WR, Hsu LL, Gordeuk VR, Viswanathan K, Sarnaik S, Osunkwo I, Guillaume E, Sadanandan S, Sieger L, Lasky JL, Panosyan EH, Blake OA, New TN, Bellevue R, Tran LT, Razon RL, Stark CW, Neumayr LD, Vichinsky EP; Investigators of the Phase 3 Trial of l-Glutamine in Sickle Cell Disease. A Phase 3 Trial of l-Glutamine in Sickle Cell Disease. N Engl J Med. 2018 Jul 19;379(3):226-235. doi: 10.1056/NEJMoa1715971. PMID 30021096

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Patients will be randomized to receive Placebo.
  Placebo (100% maltodextrin): 0.3 g/kg of placebo will be administered twice a day orally to each patient for 48 weeks. The dosage will be in increments of 5 grams based on weight. The upper limit for daily dose of study medication will be set at 30 grams. Patients will be given verbal and written instructions for self-administration of the study medication at the Baseline visit. The powder can be mixed with water or most non-heated beverages other than alcohol, or can be mixed with most non-heated foods such as yogurt, applesauce, or cereal for administration.
Period: Overall Study
Arm/Group | L-glutamine | Placebo
Started | 152 | 78
Completed | 97 | 59
Not Completed | 55 | 19

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Patients will be randomized to receive Placebo.
  Placebo: 0.3 g/kg of placebo (100% maltodextrin) will be administered twice a day orally to each patient for 48 weeks. The dosage will be in increments of 5 grams based on weight. The upper limit for daily dose of study medication will be set at 30 grams. Patients will be given verbal and written instructions for self-administration of the study medication at the Baseline visit. The powder can be mixed with water or most non-heated beverages other than alcohol, or can be mixed with most non-heated foods such as yogurt, applesauce, or cereal for administration.
- Total: Total of all reporting groups
Arm/Group | L-glutamine | Placebo | Total
Number analyzed (Participants) | 152 | 78 | 230
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 75 | 43 | 118
  Between 18 and 65 years | 77 | 35 | 112
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.4 (12.32) | 21.4 (12.42) | 22.0 (12.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 45 | 124
  Male | 73 | 33 | 106
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 144 | 73 | 217
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 8 | 5 | 13
Diagnosis [Count of Participants; unit: Participants]
  Sickle Cell Anemia | 136 | 71 | 207
  Sickle Beta plus Thalassemia | 2 | 0 | 2
  Sickle Beta zero Thalassemia | 14 | 7 | 21

OUTCOME MEASURES:

1. Primary Outcome: The Number of Occurrences of Sickle Cell Crises
Description: The number of occurrences of protocol-defined sickle cell crises that occur from Week 0 to Week 48 will be used to evaluate the efficacy of oral L-glutamine as a treatment for sickle cell anemia and beta-0 thalassemia.
Time Frame: 48 weeks
Population: Intent-to-Treat Population - Included all patients who were randomized and dispensed study medication.
Measure: Median (Full Range); unit: Number of crises
Groups:
- 100% Maltodextrin: Patients will be randomized to receive Placebo.
  100% maltodextrin: 0.3 g/kg of placebo (100% maltodextrin) will be administered twice a day orally to each patient for 48 weeks. The dosage will be in increments of 5 grams based on weight. The upper limit for daily dose of study medication will be set at 30 grams. Patients will be given verbal and written instructions for self-administration of the study medication at the Baseline visit. The powder can be mixed with water or most non-heated beverages other than alcohol, or can be mixed with most non-heated foods such as yogurt, applesauce, or cereal for administration.
Arm/Group | L-glutamine | 100% Maltodextrin
Number analyzed (Participants) | 152 | 78
Number of crises | 3 [0 to 15] | 4 [0 to 15]
Statistical Analysis 1: Comparison: L-glutamine vs 100% Maltodextrin; Test type: Superiority or Other; p = 0.0052, Cochran-Mantel-Haenszel — 1. The primary analysis was analyzed using a CMH analysis of the number of SCCs using modified ridit scores. 2. P-value (controlling for region and HU use) 3. The null hypothesis of the final analysis was performed at the 0.045 significance level; Wilcoxon rank-sum test = 0.5

2. Secondary Outcome: The Number of Hospitalizations for Sickle Cell Pain
Description: The number of hospitalizations that occur from Week 0 to Week 48, will be used to evaluate the efficacy of oral L-glutamine as a treatment for sickle cell anemia and beta-0 thalassemia.
Time Frame: 48 weeks
Population: Intent-to-Treat Population - Included all patients who were randomized and dispensed study medication.
Measure: Median (Full Range); unit: Number of hospitalizations
Arm/Group | L-glutamine | 100% Maltodextrin
Number analyzed (Participants) | 152 | 78
Number of hospitalizations | 2 [0 to 14] | 3 [0 to 13]
Statistical Analysis 1: Comparison: L-glutamine vs 100% Maltodextrin; Test type: Superiority or Other; p = 0.0045, Cochran-Mantel-Haenszel

3. Secondary Outcome: The Number of Emergency Room/Medical Facility Visits for Sickle Cell Pain
Description: The number of emergency room visits or medical facility visits that occur from Week 0 to Week 48, will be used to evaluate the efficacy of oral L-glutamine as a treatment for sickle cell anemia and beta-0 thalassemia.
Time Frame: 48 weeks
Population: Intent-to-Treat Population - Included all patients who were randomized and dispensed study medication.
Measure: Median (Full Range); unit: Number of ER visits
Arm/Group | L-glutamine | 100% Maltodextrin
Number analyzed (Participants) | 152 | 78
Number of ER visits | 1 [0 to 12] | 1 [0 to 15]
Statistical Analysis 1: Comparison: L-glutamine vs 100% Maltodextrin; Test type: Superiority or Other; p = 0.0888, Cochran-Mantel-Haenszel

4. Secondary Outcome: The Effect of Oral -L-glutamine on Hematological Parameters
Description: To assess the effect of oral L-glutamine on hematological parameters (hemoglobin), Change from Baseline will be reported at Weeks 4, 24 and 48.
Time Frame: Baseline, Week 4, 24 and 48
Population: Safety population - The safety population included all patients who received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | L-glutamine | Placebo
Number analyzed (Participants) | 151 | 78
g/dL
  Hemoglobin at Baseline | 8.82 (1.43) | 8.71 (1.17)
  Change in Hemoglobin at week 4: number analyzed (Participants) | 134 | 69
  Change in Hemoglobin at week 4 | 0.04 (0.84) | 0.23 (0.71)
  Change in Hemoglobin at Week 24: number analyzed (Participants) | 99 | 61
  Change in Hemoglobin at Week 24 | -0.17 (1.01) | -0.12 (1.24)
  Change in Hemoglobin at Week 48: number analyzed (Participants) | 80 | 47
  Change in Hemoglobin at Week 48 | -0.12 (0.95) | -0.12 (0.96)

5. Secondary Outcome: The Effect of Oral L-glutamine on Vital Signs
Description: To assess the effect of oral L-glutamine on Vital signs (systolic and diastolic blood pressure). Change from Baseline will be reported at Weeks 4, 24, and 48.
Time Frame: Baseline, Week 4, 24, and 48
Population: Safety Population which includes all patients that took at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | L-glutamine | 100% Maltodextrin
Number analyzed (Participants) | 151 | 78
mm Hg
  Systolic blood pressure at Baseline | 111.3 (11.20) | 114.6 (14.16)
  Change Systolic blood pressure at Week 4: number analyzed (Participants) | 134 | 73
  Change Systolic blood pressure at Week 4 | 0.5 (11.19) | -0.2 (10.68)
  Change in Systolic blood pressure at Week 24: number analyzed (Participants) | 102 | 63
  Change in Systolic blood pressure at Week 24 | 1.1 (10.78) | 0.5 (14.23)
  Change in Systolic blood pressure at Week 48: number analyzed (Participants) | 86 | 51
  Change in Systolic blood pressure at Week 48 | 2.2 (10.78) | 2.6 (15.70)
  Diastolic blood pressure at Baseline | 64.8 (8.61) | 66.2 (9.75)
  Change in Diastolic blood pressure at Week 4: number analyzed (Participants) | 134 | 73
  Change in Diastolic blood pressure at Week 4 | -0.7 (9.08) | 0.3 (10.29)
  Change in Diastolic blood pressure at Week 24: number analyzed (Participants) | 102 | 63
  Change in Diastolic blood pressure at Week 24 | -0.7 (8.40) | 0.6 (12.44)
  Change in Diastolic blood pressure at Week 48: number analyzed (Participants) | 86 | 51
  Change in Diastolic blood pressure at Week 48 | 0.4 (8.71) | 2.0 (9.96)

6. Secondary Outcome: The Effect of Oral L-glutamine on Hematological Parameters
Description: To assess the effect of oral L-glutamine on hematological parameters (hematocrit), Change from Baseline will be reported at Weeks 4, 24 and 48.
Time Frame: Baseline, Week 4, 24 and 48
Population: Safety population - The safety population included all patients who received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: % of red blood cells
Arm/Group | L-glutamine | 100% Maltodextrin
Number analyzed (Participants) | 151 | 78
% of red blood cells
  Hematocrit at Baseline | 27.67 (4.40) | 27.53 (3.61)
  Change in Hematocrit at Week 4 | 0.16 (2.77) | 0.75 (2.52)
  Change in Hematocrit Week 24 | -0.26 (3.42) | -0.15 (4.13)
  Change in Hematocrit at Week 48 | 0.16 (3.27) | 0.11 (3.19)

7. Secondary Outcome: The Effect of Oral L-glutamine on Hematological Parameters
Description: To assess the effect of oral L-glutamine on hematological parameters (reticulocyte count), Change from Baseline will be reported at Weeks 4, 24 and 48.
Time Frame: Baseline, Week 4, 24 and 48
Population: Safety population - The safety population included all patients who received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: 1000 cells/uL
Arm/Group | L-glutamine | 100% Maltodextrin
Number analyzed (Participants) | 151 | 78
1000 cells/uL
  Reticulocyte (Abs) | 283.62 (129.49) | 295.03 (140.10)
  Change in Reticulocyte (Abs) at Week 4 | -9.28 (104.88) | -23.09 (160.41)
  Change in Reticulocyte (Abs) at Week 24 | 7.94 (111.85) | -1.93 (137.65)
  Change in Reticulocyte (Abs) at Week 48 | 50.89 (112.93) | 26.27 (140.65)

8. Secondary Outcome: The Effect of Oral L-glutamine on Vital Signs
Description: To assess the effect of oral L-glutamine on Vital signs (pulse rate). Change from Baseline will be reported at Weeks 4, 24, and 48.
Time Frame: Baseline, Week 4, Week 24 and Week 48
Population: Safety Population which includes all patients that took at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | L-glutamine | 100% Maltodextrin
Number analyzed (Participants) | 151 | 78
bpm
  Pulse Rate (bpm) at Baseline | 85.6 (13.15) | 88.5 (14.07)
  Change in Pulse Rate (bpm) at Week 4: number analyzed (Participants) | 134 | 73
  Change in Pulse Rate (bpm) at Week 4 | -0.1 (12.07) | -0.4 (14.96)
  Change in Pulse Rate (bpm) at Week 24: number analyzed (Participants) | 102 | 63
  Change in Pulse Rate (bpm) at Week 24 | 3.0 (14.58) | -1.5 (15.05)
  Change in Pulse Rate (bpm) at 48: number analyzed (Participants) | 86 | 51
  Change in Pulse Rate (bpm) at 48 | 1.1 (14.74) | 0.2 (15.33)

9. Secondary Outcome: Effect of Oral L-glutamine on Vital Signs
Description: To assess the effect of oral L-glutamine on Vital signs (temperature). Change from Baseline will be reported at Weeks 4, 24, and 48.
Time Frame: Baseline, Week 4, Week 24 and Week 48
Population: Safety Population which includes all patients that took at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: degree C
Arm/Group | L-glutamine | 100% Maltodextrin
Number analyzed (Participants) | 151 | 78
degree C
  Temperature at Baseline | 36.85 (0.387) | 36.83 (0.403)
  Change in Temperature at Week 4: number analyzed (Participants) | 135 | 73
  Change in Temperature at Week 4 | -0.06 (0.436) | -0.02 (0.540)
  Change in Temperature at Week 24: number analyzed (Participants) | 102 | 63
  Change in Temperature at Week 24 | -0.05 (0.469) | 0.03 (0.510)
  Change in Temperature at Week 48: number analyzed (Participants) | 86 | 51
  Change in Temperature at Week 48 | -0.09 (0.442) | 0.05 (0.521)

10. Secondary Outcome: The Effect of Oral L-glutamine on Vital Signs
Description: To assess the effect of oral L-glutamine on Vital signs (respiration). Change from Baseline will be reported at Weeks 4, 24, and 48.
Time Frame: Baseline, Week 4, Week 24 and Week 48
Population: Safety Population which includes all patients that took at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: breaths/min
Arm/Group | L-glutamine | 100% Maltodextrin
Number analyzed (Participants) | 151 | 78
breaths/min
  Respiration at Baseline | 18.9 (3.0) | 19.1 (2.34)
  Change in Respiration at Week 4: number analyzed (Participants) | 133 | 73
  Change in Respiration at Week 4 | -0.2 (3.01) | -0.2 (2.55)
  Change in Respiration at Week 24: number analyzed (Participants) | 101 | 63
  Change in Respiration at Week 24 | -0.7 (3.03) | -0.6 (3.36)
  Change in Respiration at Week 48: number analyzed (Participants) | 85 | 51
  Change in Respiration at Week 48 | -0.7 (3.25) | -0.6 (2.94)

ADVERSE EVENTS:
Time Frame: Adverse events data were collected throughout the course of the study (53 weeks or about 1 year).
Description: The Safety population will include all patients who received at least one dose of study medication.
Arm/Group | L-glutamine | 100% Maltodextrin
Serious Adverse Events (participants affected / at risk) | 118/151 | 68/78
Other Adverse Events (participants affected / at risk) | 148/151 | 78/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | L-glutamine (N=151) | 100% Maltodextrin (N=78)
Acute Chest Syndrome (Blood and lymphatic system disorders) | 12 | 18
Anaemia (Blood and lymphatic system disorders) | 1 | 2
Aplastic anaemia (Blood and lymphatic system disorders) | 1 | 0
Haemolysis (Blood and lymphatic system disorders) | 1 | 0
Hypersplenism (Blood and lymphatic system disorders) | 2 | 0
Leucocytosis (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0
Cardiac Arrest (Cardiac disorders) | 2 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Sickle cell anaemia with crisis (Congenital, familial and genetic disorders) | 102 | 63
Eye irritation (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 3
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1
Gastritis (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Pancreatic acute (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 1
Chest pain (General disorders) | 5 | 1
Death (General disorders) | 1 | 0
Drug withdrawal syndrome (General disorders) | 0 | 1
Necrosis (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 2 | 0
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 6 | 3
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (General disorders) | 1 | 0
Hyperbilirubinaemia (General disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 1
Gastroenteritis (Infections and infestations) | 0 | 2
Gastrointestinal viral infection (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 3 | 1
Lobar pneumonia (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 0
Osteomyelitis acute (Infections and infestations) | 0 | 1
Pharnygitis streptococcal (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 3 | 8
Sepsis (Infections and infestations) | 1 | 0
Sinustitis (Infections and infestations) | 1 | 1
Tonsilitis (Infections and infestations) | 0 | 1
Tooth infection (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Complication of device removal (Injury, poisoning and procedural complications) | 1 | 0
Device leakage (Injury, poisoning and procedural complications) | 0 | 1
Device malfunction (Injury, poisoning and procedural complications) | 2 | 0
Device occlusion (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Haemolytic transfusion reaction (Injury, poisoning and procedural complications) | 1 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 1
Post-traumatic reaction (Injury, poisoning and procedural complications) | 1 | 0
Traumatic arthropathy (Injury, poisoning and procedural complications) | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1
White blood cell count increased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 2
Hyperkalaemia (Investigations) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Bunion (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone infarction (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0
Dysarthria (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 1
Migraine (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 2 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 2 | 2
Mental status changes (Psychiatric disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 1
Priapism (Reproductive system and breast disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 | 0
Hip arthroplasty (Surgical and medical procedures) | 0 | 1
Strabismus correction (Surgical and medical procedures) | 1 | 0
Tonsillectomy (Surgical and medical procedures) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 2 | 0
Thrombophlebits superficial (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | L-glutamine (N=151) | 100% Maltodextrin (N=78)
Acute chest syndrome (Blood and lymphatic system disorders) | 18 | 21
Leukocytosis (Blood and lymphatic system disorders) | 9 | 6
Anaemia (Blood and lymphatic system disorders) | 7 | 6
Tachycardia (Cardiac disorders) | 8 | 4
Sickle cell anaemia with crisis (Congenital, familial and genetic disorders) | 123 | 71
Ocular icterus (Eye disorders) | 15 | 9
Constipation (Gastrointestinal disorders) | 38 | 19
Nausea (Gastrointestinal disorders) | 34 | 13
Vomiting (Gastrointestinal disorders) | 22 | 10
Abdominal pain (Gastrointestinal disorders) | 18 | 10
Abdominal pain upper (Gastrointestinal disorders) | 16 | 6
Diarrhoea (Gastrointestinal disorders) | 12 | 5
Pyrexia (General disorders) | 33 | 29
Chest pain (General disorders) | 21 | 7
Fatigue (General disorders) | 9 | 1
Oedema peripheral (General disorders) | 8 | 8
Upper respiratory tract infection (Infections and infestations) | 27 | 18
Nasopharyngitis (Infections and infestations) | 10 | 6
Urinary tract infection (Infections and infestations) | 10 | 3
Pneumonia (Infections and infestations) | 9 | 14
Bronchitis (Infections and infestations) | 5 | 4
Gastroenteritis (Infections and infestations) | 5 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 6 | 5
Hypomanesaemia (Investigations) | 6 | 4
Hyperkalaemia (Metabolism and nutrition disorders) | 5 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 24 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 20 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 19 | 10
Headache (Nervous system disorders) | 32 | 14
Dizziness (Nervous system disorders) | 8 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 26 | 14
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 11 | 5
Oropharnyngeal pain (Respiratory, thoracic and mediastinal disorders) | 11 | 11
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 7
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 14 | 11
Rash (Skin and subcutaneous tissue disorders) | 3 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI agrees that any INFORMATION submitted to it by EMMAUS shall be maintained in secrecy for a period of seven (7) years from each disclosure of INFORMATION. PI will use the up most due diligence to prevent disclosure by it except to its employees, agents, and contractors necessary for evaluation, all of whom shall be bound by similar written obligations of confidentiality, and who agree not to use the INFORMATION for any purpose other than for evaluation purposes.